CLINICAL TRIAL: NCT00796003
Title: A Phase I/II Clinical Study of JNJ-30979754 (Decitabine) in Patients With Myelodysplastic Syndrome
Brief Title: A Study of JNJ-30979754 (Decitabine) in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015406; 30979754-JPN-MDS-101 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome; MDS; Decitabine; JNJ-30979754
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I: JNJ-30979754 15 mg/m2 (Experimental): JNJ-30979754 (decitabine) 15 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1
  Interventions: Drug: JNJ-30979754 15 mg/m2
- Phase I: JNJ-30979754 20 mg/m2 (Experimental): JNJ-30979754 (decitabine) 20 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1
  Interventions: Drug: JNJ-30979754 20 mg/m2
- Phase II: JNJ-30979754 20 mg/m2 (Experimental): JNJ-30979754 (decitabine) 20 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) cycles
  Interventions: Drug: JNJ-30979754 20 mg/m2

INTERVENTIONS:
Drug: JNJ-30979754 15 mg/m2 — JNJ-30979754 (decitabine) 15 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1.
  Other Names: decitabine
  Arms: Phase I: JNJ-30979754 15 mg/m2
Drug: JNJ-30979754 20 mg/m2 — Phase I: JNJ-30979754 (decitabine) 20 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1. Phase II: JNJ-30979754 (decitabine) 20 mg/m2 will be administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) cycles until the decitabine was expected to be effective in participants.
  Other Names: decitabine
  Arms: Phase I: JNJ-30979754 20 mg/m2; Phase II: JNJ-30979754 20 mg/m2

SUMMARY:
The purpose of this study is to to determine the recommended dose level of JNJ-30979754 (decitabine) as well as to assess the safety and effectiveness in patients with Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
This is an open-label (both physician and patient know the name and dosage of drug), multi-center study. This study consists of two parts, Phase I and Phase II. In Phase I, approximately 9 participants will be enrolled ie, 3 participants for dose level 1 (15 mg/m2 of JNJ-30979754) and 6 participants for dose level 2 (20 mg/m2 of JNJ-30979754). Once the tolerability of 20 mg/m2 is confirmed additional 30 participants will be included to receive 20 mg/m2 and approximate total participants in Phase II will be 36. This study will include screening period (within 14 days prior to the day of initial administration of Cycle 1) and dosing period (1 cycle consists of administration of study medication for first 5 consecutive days + rested for 23 days; ie, total 28 days). Cycles will be reapeated in participants in whom decitabine was expected to be effective. Safety evaluations will include assessment of adverse events, vital signs, body weight, clinical laboratory tests: hematology, blood biochemistry and urinalysis, cardiopulmonary function tests: ECG, chest X ray and oximeter analysis.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome (de novo or secondary) fitting any of the recognized French-American-British classifications: refractory anemia, refractory anemia with ringed sideroblasts, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, chronic myelomonocytic leukemia with white blood cells less than 13,000 /mm3
* International Prognostic Scoring System (IPSS) greater than or equal to 0.5 (Intermediate-1, Intermediate-2 or high risk) by bone marrow assessment and bone marrow cytogenetics within 28 days before study registration
* 20 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Normal renal and hepatic function

Exclusion Criteria:

* Acute Myeloid Leukemia (AML) with bone marrow blasts greater than or equal to 30%
* Participants with a history of high-dose cytarabine (Ara-C) therapy (greater than 1,000 mg/m2/day)
* Participants administered adrenal cortex hormones or anabolic hormones within 7 days of study initiation
* Participants who have received a colony stimulating factor (CSF) formulation within 7 days of study initiation
* Active double cancer
* Uncontrolled cardiac disease or cognitive heart failure
* Uncontrolled restrictive or obstructive pulmonary disease
* Uncontrolled diabetes mellitus
* Active viral or bacterial infection
* Known positive serology for Human immunodeficiency virus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (7):
- Japan (7):
  - Fukuoka
  - Hamamatsu
  - Hidaka
  - Nagasaki
  - Nagoya
  - Shinjuku
  - Tokyo

REFERENCES:
- [Derived] Oki Y, Kondo Y, Yamamoto K, Ogura M, Kasai M, Kobayashi Y, Watanabe T, Uike N, Ohyashiki K, Okamoto S, Ohnishi K, Tomita A, Miyazaki Y, Tohyama K, Mukai HY, Hotta T, Tomonaga M. Phase I/II study of decitabine in patients with myelodysplastic syndrome: a multi-center study in Japan. Cancer Sci. 2012 Oct;103(10):1839-47. doi: 10.1111/j.1349-7006.2012.02386.x. Epub 2012 Sep 14. PMID 22816487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 participants were enrolled at multiple sites in Japan.
Pre-assignment Details: 9 participants were enrolled and treated in Phase 1. 36 participants (including 6 participants from Phase I) were enrolled in Phase II. 34 participants were treated and 2 participants were untreated in Phase II.
Groups:
- Phase I: 15 mg/m2: 15 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of a 4-Week (28-day) Cycle 1
- Phase I and II: 20 mg/m2: Phase I: 20 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of a 4-Week (28-day) Cycle 1. Phase II: 20 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) other cycles (except Cycle I)
Period: Overall Study
Arm/Group | Phase I: 15 mg/m2 | Phase I and II: 20 mg/m2
Started | 3 (Number of participants enrolled) | 36 (Number of participants enrolled. Includes 6 participants from Phase I (20 mg/m2) group)
Treated | 3 (Number of participants treated) | 34 (Number of participants treated)
Completed | 0 | 7 (Includes 2 participants from Phase I (20 mg/m2) group)
Not Completed | 3 | 29
Not completed — Disease Progression | 2 | 13
Not completed — Adverse Event | 1 | 7
Not completed — Specified organ function not met | 0 | 1
Not completed — Physician Decision | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1
Not completed — Participants Not treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: For Baseline characteristics analysis, number of participants treated were analyzed (37) instead of number of participants enrolled (39). 2 enrolled participants were not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 15 mg/m2 | Phase I and II: 20 mg/m2 | Total
Number analyzed (Participants) | 3 | 34 | 37
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (2.08) [67 to 71] | 68.5 (7.09) | 68.5 (6.81)
Age, Customized [Number; unit: Participants]
  <65 years | 0 | 10 | 10
  >= 65 and <= 74 years | 3 | 17 | 20
  >=75 years | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 3 | 26 | 29

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Overall Remission Rate (ORR): Number of Participants Who Achieved Complete Remission (CR)+Partial Remission (PR) - as Per International Working Group (IWG) Response Criteria (2000)
Description: IWG response criteria (2000) - CR: bone marrow evaluations show < 5% blasts; no dysplasia; normal maturation of all cell lines and peripheral blood shows hemoglobin ≥ 11 g/dL; neutrophils ≥ 1,500/mL; platelets ≥ 100,000/mL; 0% blasts; no dysplasia and PR: same as CR, except blasts decrease by ≥ 50% or lower French-American-British (FAB) classification of Myelodysplastic Syndromes.
Time Frame: Up to 1 years after the last participant enrolled
Population: Full Analysis Set (FAS): 34 participants were included in this analysis set for Phase II
Measure: Number; unit: Participants
Groups:
- Phase II: 20 mg/m2: 20 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) cycles
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 34
Participants
  CR | 7
  PR | 2
Statistical Analysis 1: Comparison: Phase II: 20 mg/m2; Null Hypothesis: Overall Remission Rate = 5%; Test type: Superiority or Other; p < 0.0001, Binomial test; one-tailed 5% level at a significance level; Overall Response Rate = 26.5, 90% CI 2-sided [14.6 to 41.6], Standard Error of Mean 7.6

2. Primary Outcome: Phase I and II: Number of Participants Who Experienced Adverse Events
Time Frame: Up to 1.5 years after the last participant enrolled
Population: Safety Population: 9 participants in Phase I and 34 participants in Phase II were evaluated for safety
Measure: Number; unit: Participants
Groups:
- Phase I: 20 mg/m2: 20 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of a 4-Week (28-day) Cycle 1
Arm/Group | Phase I: 15 mg/m2 | Phase I: 20 mg/m2 | Phase II: 20 mg/m2
Number analyzed (Participants) | 3 | 6 | 34
Participants | 3 | 6 | 34

3. Secondary Outcome: Phase I: Maximum Observed Plasma Concentration of Decitabine (Cmax)
Time Frame: Before dosing (Pre-dose), 30 min, 60 min (end of infusion), 65 min, 75 min, 90 min, 120 min, 180 min, 240 min after the start of decitabine infusion on Day 1 and Day 5 of 28-Days Cycle 1
Population: Pharmacokinetic Population: 8 participants were evaluated for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I: 15 mg/m2 | Phase I: 20 mg/m2
Number analyzed (Participants) | 3 | 5
ng/mL
  Day 1 | 151.7 (28.729) | 166.4 (17.170)
  Day 5 | 142.0 (40.635) | 190.6 (54.679)

4. Secondary Outcome: Phase I: Area Under the Plasma Concentration-time Curve (AUC)
Description: Area under the curve from time zero to extrapolated infinite time (AUC Infinity) and area under the curve from time zero to last quantifiable concentration (AUC Last).
Time Frame: as for outcome 3
Population: Pharmacokinetic Population: 8 participants were evaluated for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase I: 15 mg/m2 | Phase I: 20 mg/m2
Number analyzed (Participants) | 3 | 5
ng*h/mL
  AUC Last - Day 1 | 149.0 (41.102) | 155.2 (15.754)
  AUC Last - Day 5 | 136.0 (37.855) | 152.0 (15.712)
  AUC Infinity - Day 1 | 150.0 (40.777) | 156.1 (15.497)
  AUC Infinity - Day 5 | 136.9 (37.897) | 151.2 (17.617)

5. Secondary Outcome: Phase I: Number of Participants Who Achieved Complete Remission (CR)+Partial Remission (PR)+Hematological Improvement (HI) - as Per International Working Group (IWG) Response Criteria (2000)
Description: IWG response criteria (2000) - CR: bone marrow evaluations (mCR) show < 5% blasts; no dysplasia; normal maturation of all cell lines and peripheral blood shows hemoglobin ≥ 11 g/dL; neutrophils ≥ 1,500/mL; platelets ≥ 100,000/mL; 0% blasts; no dysplasia; PR: same as CR, except blasts decrease by ≥ 50% or lower French-American-British (FAB) classification of Myelodysplastic Syndromes; HI: hemoglobin < 11 g/dL (erythroid); platelet < 100,000/mL; neutrophils < 1,000/mL.
Time Frame: Up to 28 Days of treatment Cycle 1
Population: Full Analysis Set (FAS): 9 participants were included in this set for Phase I
Measure: Number; unit: Participants
Arm/Group | Phase I: 15 mg/m2 | Phase I: 20 mg/m2
Number analyzed (Participants) | 3 | 6
Participants
  PR | 1 | 1
  HI | 1 | 2

6. Secondary Outcome: Phase II: Median Time to Remission
Description: Median time required for the participants to achieve remission (complete remission+partial remission).
Time Frame: Up to 1.5 years after the last participant enrolled
Population: 9 participants who achieved remission were evaluated.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 9
Days | 130.0 [67.0 to 208.0]

7. Secondary Outcome: Phase II: Median Time to Improvement
Description: Median time required for the participants to achieve overall improvement (complete remission+partial remission+hematologic improvement)
Time Frame: Up to 1.5 years after the last participant enrolled
Population: 14 participants who achieved overall improvement were evaluated.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 14
Days | 26.5 [22.0 to 36.0]

8. Secondary Outcome: Phase II: Median Duration of Remission
Description: Median time duration for which participants achieved remission (complete remission+partial remission).
Time Frame: Up to 1.5 years after the last participant enrolled
Population: 9 participants who achieved remission were evaluated.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 9
Days | 489 [294 to 489]

9. Secondary Outcome: Phase II: Median Duration of Overall Improvement
Description: Median time duration for which participants achieved overall improvement (complete remission+partial remission+hematologic improvement).
Time Frame: Up to 1.5 years after the last participant enrolled
Population: 14 participants who achieved overall improvement were evaluated.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 14
Days | 532 [147 to 554]

10. Secondary Outcome: Phase II: Overall Improvement Rate: Number of Participants Who Achieved Complete Response (CR)+Partial Response (PR)+Hematological Improvement (HI) - as Per International Working Group (IWG) Response Criteria (2000)
Description: IWG response criteria (2000) - CR: bone marrow evaluations (mCR) show < 5% blasts; no dysplasia; normal maturation of all cell lines and peripheral blood shows hemoglobin ≥ 11 g/dL; neutrophils ≥ 1,500/mL; platelets ≥ 100,000/mL; 0% blasts; no dysplasia and PR: same as CR, except blasts decrease by ≥ 50% or lower French-American-British (FAB) classification of Myelodysplastic Syndromes. HI: hemoglobin < 11 g/dL (erythroid); platelet < 100,000/mL; neutrophils < 1,000/mL.
Time Frame: Up to 1.5 years after the last participant enrolled
Population: Full Analysis Set (FAS): 34 participants were included in this set
Measure: Number; unit: Participants
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 34
Participants
  CR | 7
  PR | 2
  HI | 5

11. Secondary Outcome: Phase II: Number of Participants With Cytogenic Response - as Per International Working Group (IWG) Response Criteria 2000 (Major/Minor) and IWG 2006 (Complete/Partial)
Description: IWG 2000 - Major: disappearance of cytogenetic abnormality; Minor: 50% or more reduction in abnormal metaphases. IWG 2006 - Complete: disappearance of the chromosomal abnormality without appearance of new ones; Partial: At least 50% reduction of the chromosomal abnormality.
Time Frame: Up to 1.5 years after the last participant enrolled
Population: 20 participants who had chromosomal abnormality were evaluated in Phase II for cytogenetic response. The IWG criteria requires 20 analyzable metaphases using conventional cytogenetic techniques.
Measure: Number; unit: Participants
Arm/Group | Phase II: 20 mg/m2
Number analyzed (Participants) | 20
Participants
  Major/Complete | 6
  Minor/Partial | 1
  No response | 10
  Not estimable | 3

ADVERSE EVENTS:
Time Frame: Up to 1.5 years after the last participant enrolled
Groups:
- Phase I - 15 mg/m2 Group: 15 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1
- Phase I - 20 mg/m2 Group: 20 mg/m2 of JNJ-30979754 (decitabine) administered once daily by 1-hour intravenous infusion from Day 1 to 5 of 4-Week (28-day) Cycle 1
Arm/Group | Phase I - 15 mg/m2 Group | Phase I - 20 mg/m2 Group | Phase II: 20 mg/m2
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 11/34
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - 15 mg/m2 Group (N=3) | Phase I - 20 mg/m2 Group (N=6) | Phase II: 20 mg/m2 (N=34)
Pneumonia (Infections and infestations) | 1 | 0 | 4
Sepsis (Infections and infestations) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Aneamia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - 15 mg/m2 Group (N=3) | Phase I - 20 mg/m2 Group (N=6) | Phase II: 20 mg/m2 (N=34)
Neutropenic infection (Infections and infestations) | 2 | 3 | 15
Pneumonia (Infections and infestations) | 0 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 6
Oral herpes (Infections and infestations) | 0 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 6 | 34
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 29
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6 | 27
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 6
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 4
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 3 | 8
Confusional state (Psychiatric disorders) | 0 | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 3
Somnolence (Nervous system disorders) | 0 | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 1 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 4
Haematoma (Vascular disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 3 | 14
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 9
Nausea (Gastrointestinal disorders) | 1 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 3
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 13
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 10
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2
Injection site reaction (General disorders) | 0 | 2 | 10
Fatigue (General disorders) | 0 | 2 | 6
Pyrexia (General disorders) | 1 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 17
Alanine aminotransferase increased (Investigations) | 1 | 1 | 15
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 14
Protein total decreased (Investigations) | 0 | 2 | 13
Blood albumin decreased (Investigations) | 0 | 2 | 12
Blood bilirubin increased (Investigations) | 1 | 1 | 11
Blood glucose increased (Investigations) | 0 | 1 | 12
Blood urine present (Investigations) | 0 | 5 | 11
Weight decreased (Investigations) | 1 | 2 | 7
Blood potassium decreased (Investigations) | 0 | 1 | 7
Blood sodium decreased (Investigations) | 0 | 1 | 6
Protein urine present (Investigations) | 0 | 1 | 5
Blood bicarbonate decreased (Investigations) | 0 | 1 | 4
Blood potassium increased (Investigations) | 0 | 0 | 4
C-reactive protein increased (Investigations) | 3 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 3
Blood urea increased (Investigations) | 0 | 1 | 3
Blood amylase increased (Investigations) | 0 | 0 | 2
Glucose urine present (Investigations) | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 1 | 11
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 4
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days